CLINICAL TRIAL: NCT07321444
Title: Effectiveness of Telerehabilitation in Shoulder Pathology
Brief Title: Telerehabilitation in Shoulder Pathology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Yolanda Marcen Roman, PhD, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.P.-C.I. PI21-403
Record Dates: First submitted 2025-09-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Pathology
Keywords: Telerehabilitation; Physiotherapy; Physical Therapy; Shoulder
MeSH Terms: interventions — Telerehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): exercises supervised by videoconference
  Interventions: Procedure: telerehabilitation in physiotherapy
- Face to face physiotherapy (Active Comparator): Face to face exercise sessions in the physiotherapy room
  Interventions: Procedure: face to face physiotherapy

INTERVENTIONS:
Procedure: telerehabilitation in physiotherapy — Exercises supervised by videoconference.
  Arms: Telerehabilitation
Procedure: face to face physiotherapy — Exercises performed in a physical therapy room.
  Arms: Face to face physiotherapy

SUMMARY:
A randomized clinical trial will be conducted to evaluate the effectiveness of telerehabilitation compared to in-person physiotherapy in the treatment of rotator cuff injuries of the shoulder. Follow-up assessments will be performed at 2, 5, and 8 weeks. Scales will be used to evaluate shoulder function, quality of life, pain perception, and satisfaction with the digital tool.

DETAILED DESCRIPTION:
Digital health is undergoing significant development in various healthcare settings, especially in primary care. Digital physiotherapy, or telerehabilitation, is a resource that promotes self-care and allows for remote monitoring and follow-up. This study focuses on its application to degenerative rotator cuff disease of the shoulder. This is justified by its high prevalence and the geographical dispersion of the population served by the Primary Care Physiotherapy Unit of Teruel Ensanche. Objectives: The main objective is to evaluate the effectiveness of a primary care telerehabilitation program for patients with degenerative rotator cuff disease of the shoulder, compared to traditional physiotherapy. Secondary objectives are to assess patients' perception and satisfaction with this intervention and to analyze the usability and acceptance of the telerehabilitation program. Methodology: A 12-week randomized clinical trial will be conducted at the Teruel Ensanche Health Center. A sample of 68 adults aged 34 to 87 years with degenerative rotator cuff disease of the shoulder was estimated. Participants require internet access and an electronic device. The variables measured: shoulder function (Constant-Murley test), degree of disability (DASH questionnaire), quality of life (COOP/WONCA questionnaire), and pain perception (numerical rating scale). The intervention group (IG) receive an individualized program with remotely guided and supervised exercises, supplemented by a weekly in-person session. The control group (CG) receive standard treatment: 10 in-person physiotherapy sessions, followed by unsupervised home exercises. Assessments will be conducte at baseline and at 2, 5, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18.
* Diagnosis of degenerative shoulder rotator cuff disease.
* Internet access.
* Access to a video calling device.

Exclusion Criteria:

* Previous shoulder surgery.
* Cognitive impairment that prevents them from performing the task.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder functionality | At baseline, at 2, 5, 8, and 12 weeks.
  Shoulder function will be analyzed using the test Constant Murley.A maximum total score of 100 indicates optimal health and mobility in this joint. The results are divided into four main categories: pain (15 points), activities of daily living (20 points), mobility (40 points), and strength (25 points). It is essential to distinguish between scores below 60, which denote a severely dysfunctional state, and those above 80, which reflect optimal functionality.

SECONDARY OUTCOMES:
Health-related quality of life | At baseline, and at 2, 5, 8, and 12 weeks.
  The COOP-WONCA questionnaire The COOP-WONCA questionnaire is a brief instrument for assessing health status and health-related quality of life (HRQoL), widely used in primary care and clinical studies to obtain a global and functional view of the patient's perceived health status.
  It consists of 7 items, and scores were processed using a 5-point Likert scale, with higher scores corresponding to a poorer quality of life.
Level of shoulder disability | At baseline, 5 and 12 weeks
  Shoulder disability will be analyzed using the DASH questionnaire (Disabilities of the Arm, Shoulder and Hand).
  The DASH consists of 30 items. Each question must be answered using a 5-point scale, where 1 indicates "No difficulty" and 5 indicates "Unable to perform." A higher score indicates greater disability.
Pain perception | At baseline, 2,5,8 and 12 weeks
  Pain perception will be analyzed using the Numerical Pain Rating Scale. It is scored from 1 to 10. The higher the score, the greater the perception of pain.
Level of satisfaction with telerehabilitation | At 12 weeks.
  Satisfaction with the use of telerehabilitation will be measured using the TUQ questionnaire (Telehealth Usability Questionnaire). It has 12 items, rated on a Likert scale from 1 to 7, the higher the score, the greater the satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Teruel Ensanche Primary Care, Teruel, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No
This study is not complete.